CLINICAL TRIAL: NCT03469635
Title: Impact of Sleeve Gastrectomy and Roux-en-Y Gastric Bypass on Fetal Growth and Relationship With the Nutritional Status of Pregnant Women
Brief Title: Nutritional Status During Pregnancy After Bariatric Surgery
Acronym: PREGNUTRIBAR
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-033
Record Dates: First submitted 2018-01-02; First posted 2018-03-19 (Actual); Last update posted 2018-03-19 (Actual); Status verified 2017-12

CONDITIONS: Nutritional Deficiency in Pregnancy (Disorder); Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Nutritional deficiencies in pregnant women after bariatric surgery — compare maternal nutritional parameters and neonatal outcomes after Roux-en-Y gastric bypass (RYGB) and sleeve gastrectomy (SG) and to assess the impact of nutritional alterations on fetal growth.

SUMMARY:
Background: There is a lack of evidence on whether maternal nutritional deficiencies after Roux-en-Y gastric bypass (RYGB) or sleeve gastrectomy (SG) affect fetal development. The investigators hypothesis is that SG could induce nutritional deficiencies during pregnancy, as RYGB does, because of food restriction. These nutritional deficiencies may alter fetal growth. Methods: Women with singleton pregnancies who had at least one nutritional evaluation during pregnancy in our institution between 2006 and 2017 were included. The investigators evaluated nutritional deficiencies according to standard and pregnancy-specific norms. They have planned to study the relationships between these parameters and fetal growth. Objectives: To compare maternal nutritional parameters and neonatal outcomes after RYGB and SG and to assess the impact of nutritional alterations on fetal growth.

DETAILED DESCRIPTION:
Design: this study is a retrospective observational study, based on a single-centre database established since 2004 at the Louis Mourier Hospital in patients who have undergone bariatric surgery. This study focuses on women who have had at least one nutritional assessment at Louis Mourier Hospital during their pregnancy between 2004 and 2017. Clinical and biological data from the database and the data from delivery collected for usual care will be used retrospectively for this study. Main objective: to compare fetal growth after SG and RYGB. Primary endpoint: measurement of birth weight.

Secondary objectives and endpoints: - to compare fetal growth after SG and RYGB adjusted for gestational age and sex (birth weight Z-score).

* to compare the number of small for gestational age after SG and RYGB (birth weight Z-score <10 th percentile)
* to compare after SG and RYGB nutritional parameters including the following evaluation criteria:

  1. Before pregnancy: weight and body mass index, weight loss between surgery and early pregnancy
  2. During pregnancy: weight gain, dietary intake, biological parameters measured in the second trimester of pregnancy, in blood (iron, ferritin, transferrin saturation, calcium, magnesium, albumin, pre-albumin, vitamins A , D, E, C, B1, B6, B9, B12, zinc, selenium, parathyroid hormone, homocysteine, hemoglobin, mean cell volume, hematocrit, blood glucose, triglycerides, cholesterol, insulin) and urine (calcium, urea, creatinine).
* to compare the number of nutritional deficiencies (number of deficiencies for each parameter listed above) after SG and RYGB with standard and pregnancy norms.
* to compare the type of deficiency after SG and RYGB (difference between the 2 types of surgery for each parameter)
* to study the relationship between nutritional parameters and fetal growth after bariatric surgery (correlations between concentrations of nutritional parameters, birth weight and birth weight Z-score)
* to study the relationship between nutritional parameters and fetal growth after each type of surgery (SG and RYGB).

Population studied: pregnant women after bariatric surgery including RYGB and SG. Practical implementation: for women who are referred to our institution during pregnancy, systematic vitamin supplementation is prescribed and then adjusted according to the nutritional dosages performed at least once a trimester. All women benefit from a systematic investigation, which includes a medical consultation, a dietary survey and fasting biological tests according to our routine post-operative evaluation. These data are prospectively collected in a database. They will be used for the study retrospectively. The birth data collected in the medical file at the end of the pregnancy will also be used for the study retrospectively. An oral agreement was obtained from all women for the collection of these data for research and a non opposition form was sended. A questionnaire was sent to women for whom there was missing data concerning their delivery.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women age > 18, who have undergone sleeve gastrectomy or Roux-en-Y gastric bypass and performed at least one nutritional evaluation during the pregnancy

Exclusion Criteria:

* twin pregnancy
* pregnant women operated by another procedure
* women who refused that data of nutritional status or delivery were used for the research

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: pregnant women after bariatric surgery
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2006-01 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
birth weight | at birth

SECONDARY OUTCOMES:
birth weight Z-score | at birth
number of newborns with birth weight Z-score < 10 th percentile | at birth
pre pregnancy weight (kg) | beginning (1st week) and end of pregnancy (39 +/- 4 weeks)
weight gain during pregnancy (kg) | end of pregnancy (39 +/- 4 weeks)
caloric intake during pregnancy (Kcal/day) | second trimester of pregnancy (between 3 and 6 months of pregnancy)
protein intake during pregnancy (g/day) | second trimester of pregnancy (between 3 and 6 months of pregnancy)
number of nutritional deficiencies during pregnancy | second trimester of pregnancy (between 3 and 6 months of pregnancy)
  nutritional parameters below the low normal value of usual norms

CONTACTS AND LOCATIONS:
Overall Officials: Muriel Coupaye, MD, Principal Investigator — Assistance Publique Hopitaux de Paris